CLINICAL TRIAL: NCT03252743
Title: Internet-delivered Exposure-based Cognitive Behavior Therapy for Pain-predominant Functional Gastrointestinal Disorders in Children and Adolescents: an Implementation Study.
Brief Title: ICBT for Pain-predominant FGIDs in Children and Adolescents: an Implementation Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marianne Bonnert, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGID IMP 2017
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Functional Gastrointestinal Disorders; Irritable Bowel Syndrome; Dyspepsia; Functional Abdominal Pain
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome; Dyspepsia

STUDY DESIGN:
Intervention Model Description: Open trial without control group to test feasibility and evaluate preliminary effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered CBT (Experimental): Exposure-based internet-delivered CBT with ten weekly modules distributed over the internet during ten weeks, and weekly therapist support over the internet.
  Interventions: Behavioral: Exposure-based internet-delivered CBT

INTERVENTIONS:
Behavioral: Exposure-based internet-delivered CBT — The main target in treatment is exposure for abdominal symptoms by reducing avoidance and provoking symptoms. Participants are encouraged to gradually increase the difficulty by combining multiple challenges.
  The parents are taught how to reduce the risk for reinforcement of children's symptom behavior, and to support their child to complete the treatment.
  All treatment content is delivered over the internet, containing texts, videos, audio-files and examples. The modules are unlocked sequentially as participants worked their way through the treatment.
  Therapist support consists primarily of encouragement of any progress made in the treatment and support to find individual exercises.

SUMMARY:
This open trial aims to evaluate feasibility and preliminary effectiveness of an internet-delivered CBT-program for children and adolescents with functional gastrointestinal disorders when implemented in regular care.

DETAILED DESCRIPTION:
Pain predominant functional gastrointestinal disorders (P-FGIDs) are common in children and adolescents and associated with impaired quality of life. Our research group have previously in a series of efficacy-studies shown that internet-delivered exposure-based CBT leads to reduced symptoms and increased quality of life in children and adolescents with P-FGIDs. There is therefore reason to investigate how the treatment should be disseminated in regular care. This open trial aim to evaluate feasibility and preliminary treatment effects in regular care of the internet-delivered CBT-program for children and adolescents with P-FGIDs.

Method: Open trial with a pretest-posttest-design and no control group. The internet-delivered CBT-program is 10 week long and include weekly therapist support, consisting of online messages and telephone calls. Assessment points are baseline, weekly during treatment, post-treatment and follow-up at 3 months and 6 months after treatment completion.

Analysis: Effect sizes and within-group differences will be calculated in an intent-to-treat analysis using Cohens' d and Student's t-test.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 at date of inclusion.
* Fulfilling Rome IV-criteria for irritable bowel syndrome, functional dyspepsia or functional abdominal pain with a written statement from patient's physician confirming a diagnosis.
* Stable psychotropic medication for at least 1 month.

Exclusion Criteria:

* concurrent serious medical conditions.
* a psychiatric diagnosis, judged to be a more important treatment target than the abdominal pain.
* on-going structured psychological treatment.
* absence from school exceeding an average of 2 days a week the last month is a cause for exclusion since high school absence demands more intensive interventions than can be offered in ICBT.
* on-going abuse or severe parental psychiatric illness in the family.
* since treatment format assumes normal reading and writing skills, pronounced language skill deficits and learning difficulties lead to exclusion from the study.
* lack of regular internet-access.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-17 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Global gastrointestinal symptoms (CSI-24: subscale 7 items on GI-symptoms). | Baseline to 10 weeks.
  Change in global gastrointestinal symptoms from baseline to 10 weeks.

SECONDARY OUTCOMES:
Pain intensity (Faces Pain rating scale) | Baseline to 10 weeks
  Change in pain intensity from baseline to 10 weeks
Pain intensity (Faces Pain rating scale) | Baseline to 5 months.
  Change in pain intensity from baseline to 3 months follow-up.
Pain intensity (Faces Pain rating scale) | Baseline to 8 months.
  Change in pain intensity from baseline to 6 months follow-up.
Global gastrointestinal symptoms (CSI-24: subscale 7 items on GI-symptoms). | Baseline to 5 months.
  Change in global gastrointestinal symptoms from baseline to 3 months follow-up.
Global gastrointestinal symptoms (CSI-24: subscale 7 items on GI-symptoms). | Baseline to 8 months.
  Change in global gastrointestinal symptoms from baseline to 6 months follow-up.
Gastrointestinal symptoms module (PedsQL Gastro) | Baseline to 10 weeks
  Change in different dimensions of gastrointestinal symptoms (e.g. pain-related symptoms, nausea, bloating) from baseline to 10 weeks.
Gastrointestinal symptoms module (PedsQL Gastro) | Baseline to 5 months.
  Change in different dimensions of gastrointestinal symptoms (e.g. pain-related symptoms, nausea, bloating) from baseline to 3 months follow up.
Gastrointestinal symptoms module (PedsQL Gastro) | Baseline to 8 months.
  Change in different dimensions of gastrointestinal symptoms (e.g. pain-related symptoms, nausea, bloating) from baseline to 6 months follow up.
Fear for symptoms (Visceral sensitivity index) | Baseline to 10 weeks.
  Change in fear for symptoms from baseline to 10 weeks.
Fear for symptoms (Visceral sensitivity index) | Baseline to 5 months.
  Change in fear for symptoms from baseline to 3 months follow-up.
Fear for symptoms (Visceral sensitivity index) | Baseline to 8 months.
  Change in fear for symptoms from baseline to 6 months follow-up.
Avoidant behavior (IBS-BRQ) | Baseline to 10 weeks
  Change in avoidant behavior from baseline to 10 weeks.
Avoidant behavior (IBS-BRQ) | Baseline to 5 months.
  Change in avoidant behavior from baseline to 3 months follow-up.
Avoidant behavior (IBS-BRQ) | Baseline to 8 months.
  Change in avoidant behavior from baseline to 6 months follow-up.
Quality of life (PedsQL) | Baseline to 10 weeks.
  Change in quality of life from baseline to 10 weeks.
Quality of life (PedsQL) | Baseline to 5 months.
  Change in quality of life from baseline to 3 months follow-up.
Quality of life (PedsQL) | Baseline to 8 months.
  Change in quality of life from baseline to 6 months follow-up.

OTHER OUTCOMES:
Parental responses to children´s symptom behavior (ARCS) | Baseline to 10 weeks.
  Change in parental responses from baseline to 10 weeks.
Parental responses to children´s symptom behavior (ARCS) | Baseline to 5 months.
  Change in parental responses from baseline to 3 months follow-up.
Parental responses to children´s symptom behavior (ARCS) | Baseline to 8 months.
  Change in parental responses from baseline to 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Bonnert, PhD, Principal Investigator — Department of Clinical Neuroscience, Karolinska Institutet, Stockholm, Sweden.
Locations (1):
- Department of Clinical Neuroscience, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Research project homepage for studies on ICBT for pediatric FGIDs (in Swedish). — http://www.ontimagen.nu/www/